CLINICAL TRIAL: NCT02155881
Title: A Multi-Center, Double-Blind, Placebo-Controlled, Two-Arm, Parallel-Group, Phase III (Registration) Study to Assess the Efficacy and Safety of Ciclesonide Nasal Spray (Omnaris®) 200 mcg Once Daily in the Treatment of the Patients With Seasonal Allergic Rhinitis (SAR) in Russia
Brief Title: Efficacy and Safety of Ciclesonide Nasal Spray in Participants With Seasonal Allergic Rhinitis (SAR) in Russia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIC-RR-001; U1111-1152-9472 (Registry Identifier: WHO)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Drug therapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciclesonide 200 mcg (Experimental): Ciclesonide 200 mcg nasal spray, 2 actuations (sprays) per nostril (50 mcg ciclesonide/actuation), daily, for 2 weeks.
  Interventions: Drug: Ciclesonide
- Placebo (Placebo Comparator): Ciclesonide placebo-matching nasal spray, 2 actuations (sprays) per nostril, daily, for 2 weeks.
  Interventions: Drug: Ciclesonide Placebo

INTERVENTIONS:
Drug: Ciclesonide — Ciclesonide nasal spray 50 mcg/actuation
  Other Names: Omnaris®
  Arms: Ciclesonide 200 mcg
Drug: Ciclesonide Placebo — Ciclesonide placebo-matching nasal spray
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the efficacy and safety of Ciclesonide Nasal Spray 200 microgram (mcg) once daily in the treatment of seasonal allergic rhinitis (SAR) in Russian participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called ciclesonide. Ciclesonide is being tested to treat allergy symptoms in people who have SAR. This study will look at improvement of allergy symptoms in Russian participants who take ciclesonide nasal spray.

The study will enroll approximately 80 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Ciclesonide nasal spray 200 mcg
* Placebo nasal spray (dummy inactive nasal spray) - this is a nasal spray that looks like the study drug but has no active ingredient.

All participants will be asked to take 2 actuations per nostril at the same time each day throughout the study, and will be asked to record the severity of their allergy symptoms twice a day in a diary.

This multi-centre trial will be conducted in Russia. The overall time to participate in this study is up to 5 weeks. Participants will make 3 visits to the clinic, and will be contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by a participant for participation in the study.
2. SAR male and female participants aged greater than or equal to (>=) 18 years (with a history of SAR of 2 years on longer). In the Investigator's judgment the SAR must have been of sufficient severity to have required treatment (either continuous or intermittent) during this period, and was expected to require treatment for the duration of the study.
3. To have a demonstrated positive skin prick test or other serologic tests to at least 1 relevant seasonal allergen. A positive skin test is generally defined as a wheal 3 mm larger than the diluents control wheal for prick testing.
4. If female less than or equal to (<=) 65 years of age, must have a negative urine pregnancy test at screening. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control:

   1. An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following study participation;
   2. Barrier method of contraception, for example (eg), condom and/or diaphragm with spermicide while participating in the study.

Exclusion Criteria:

1. Nasal pathology, including nasal polyps, clinically relevant respiratory tract malformations, recent nasal biopsy (within 60 days), nasal trauma, nasal surgery, atrophic rhinitis, rhinitis medicamentosa (within 60 days), vasomotor rhinitis.
2. Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit AND use of a stable (maintenance) dose (30 days more) may be considered for inclusion.
3. Hypersensitivity to corticosteroid or any of the excipients in the formulation of ciclesonide.
4. A history of respiratory tract infection or disorder within 2 weeks of the screening visit or had a respiratory tract infection during baseline.
5. Presence of ocular herpes simplex or cataracts or a history of glaucoma.
6. Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta (β)-agonists; intermittent use of β-agonists is acceptable.
7. Use of intranasal immunosuppressive drugs for 30 days before Baseline.
8. Female participant who is pregnant or lactating.
9. Participation in any investigational drug trial within the 30 days preceding the Screening Visit or planned participation in another investigational drug trial at any time during this trial.
10. History of a positive test for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
11. History of alcohol or drug abuse within the preceding two years.
12. Use of any prohibited concomitant medications within the prescribed (per protocol) time spent last dose period to the Screening Visit (Visit 0) and during entire treatment duration.
13. Any condition that, in the judgment of the investigator, can be clinically significant and/or affect the participant's ability to participate in the clinical trial.
14. Exposure to systemic corticosteroids for any indication, chronic or intermittent (e.g.: contact dermatitis), during the past 2 months, or presence of an underlying condition that can reasonably be expected to require treatment with corticosteroids during the course of the study.
15. Use of topical corticosteroids in concentrations in excess of 1 percent (%) hydrocortisone for dermatological conditions during the past 1 month, or presence of an underlying condition that can reasonably be expected to require treatment with such preparations during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (5):
- Russia (5):
  - Kazan'
  - Krasnodar
  - Moscow
  - Saratov
  - Stavropol

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in Russia from 12 August 2014 to 14 November 2014.
Pre-assignment Details: Participants with a historical diagnosis of seasonal allergic rhinitis (SAR) were enrolled in 1 of 2 treatment groups as follows: Ciclesonide 200 microgram (mcg) and Placebo.
Groups:
- Ciclesonide 200 mcg: Ciclesonide 200 mcg, 2 puffs per nostril (50 mcg/puff), nasal spray, once daily for up to 14 days.
- Placebo: Ciclesonide placebo-matching puffs, 2 puffs per nostril, nasal spray, once daily for up to 14 days.
Period: Overall Study
Arm/Group | Ciclesonide 200 mcg | Placebo
Started | 40 | 40
Completed | 38 | 36
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Inappropriately randomized | 2 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of double-blind study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide 200 mcg | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.98 (13.16) | 38.55 (11.94) | 39.76 (12.55)
Gender [Count of Participants; unit: Participants]
  Female | 28 | 17 | 45
  Male | 12 | 23 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  White | 40 | 40 | 80
Region of Enrollment [Number; unit: participants]
  Russia | 40 | 40 | 80
Smoking Status [Number; unit: participants]
  Current Smoker | 2 | 1 | 3
  Ex-Smoker | 1 | 5 | 6
  Had Never Smoked | 37 | 34 | 71
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 70.03 (16.69) | 72.51 (16.81) | 71.27 (16.75)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.45 (10.87) | 171.45 (7.45) | 168.95 (9.16)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Over 2 Weeks in Participant-Reported Morning and Evening Reflective Total Nasal Symptom Scores (TNSS)
Description: The reflective TNSS is defined as the sum of the participant-rated reflective symptom scores for the 4 nasal symptoms of runny nose, itchy nose, sneezing, and nasal congestion over the past 12 hours. Each symptom was evaluated by the participant in an assessment diary, once in the morning (AM score) and after 12 hours in the evening (PM score) over 2 weeks of treatment period and was rated on a severity scale ranging from 0 to 3, where: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe (symptom hard to tolerate, interferes with daily activities/sleeping). TNSS score ranges from 0-12 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. The baseline value was defined as the average score over the Day -6 to Day 0. Change from Baseline was thus calculated as the 2-week average score recorded from Day 1 up to Day 14 minus the Baseline score.
Time Frame: Baseline and Week 1 up to Week 2 (entire treatment period)
Population: FAS included all randomized participants who received at least 1 dose of double-blind study medication and who had 1 baseline and at least 1 post-baseline value. Missing data was imputed using Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ciclesonide 200 mcg | Placebo
Number analyzed (Participants) | 40 | 40
scores on a scale
  Baseline | 7.81 (1.83) | 7.71 (1.63)
  Change Over 2 Weeks | -2.85 (2.47) | -2.68 (2.11)
Statistical Analysis 1: Comparison: Ciclesonide 200 mcg vs Placebo; An analysis of covariance (ANCOVA) model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.9716, ANCOVA; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.98 to 1.01]

2. Secondary Outcome: Change From Baseline Over 2 Weeks in Participant-Reported Morning and Evening Instantaneous Total Nasal Symptom Scores
Description: The instantaneous TNSS is defined as the sum of the participant-rated instantaneous symptom scores for the 4 nasal symptoms of runny nose, itchy nose, sneezing, and nasal congestion at the time of evaluation. Each symptom was evaluated by the participant in an assessment diary, once in the morning (AM score) and after 12 hours in the evening (PM score) over 2 weeks of treatment period and was rated on a severity scale ranging from 0 to 3, where: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe (symptom hard to tolerate, interferes with daily activities/sleeping). TNSS score ranges from 0-12 with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms. The baseline value was defined as the average score over the Day -6 to Day 0. Change from Baseline was thus calculated as the 2-week average score recorded from Day 1 up to Day 14 minus the Baseline score.
Time Frame: Baseline and Week 1 up to Week 2 (entire treatment period)
Population: FAS included all randomized participants who received at least 1 dose of double-blind study medication and who had 1 baseline and at least 1 post-baseline value. Missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ciclesonide 200 mcg | Placebo
Number analyzed (Participants) | 40 | 40
scores on a scale
  Baseline | 7.81 (1.85) | 7.64 (1.90)
  Change Over 2 Weeks | -2.76 (2.34) | -2.62 (2.10)
Statistical Analysis 1: Comparison: Ciclesonide 200 mcg vs Placebo; An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.8713, ANCOVA; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.87 to 1.02]

3. Secondary Outcome: Change From Baseline Over 2 Weeks in Participant-Reported Morning and Evening Reflective Total Ocular Symptom Scores (TOSS)
Description: The reflective TOSS is defined as the sum of the participant-rated reflective symptom scores for 3 ocular symptoms of itching/burning eyes, tearing/watering eyes, and redness of eyes over the past 12 hours. Each symptom was evaluated by the participant in an assessment diary, once in the morning (AM score) and after 12 hours in the evening (PM score) over 2 weeks of treatment period and was rated on a severity scale ranging from 0 to 3, where: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe (symptom hard to tolerate, interferes with daily activities/sleeping). Reflective TOSS score ranges from 0-9 with 0 representing an absence of symptoms and 9 representing severe symptoms. The baseline value was defined as the average score over the Day -6 to Day 0. Change from Baseline was thus calculated as the 2-week average score recorded from Day 1 up to Day 14 minus the Baseline score.
Time Frame: Baseline and Week 1 up to Week 2 (entire treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ciclesonide 200 mcg | Placebo
Number analyzed (Participants) | 40 | 40
scores on a scale
  Baseline | 4.78 (1.20) | 4.75 (1.32)
  Change Over 2 Weeks | -1.68 (1.66) | -1.68 (1.66)
Statistical Analysis 1: Comparison: Ciclesonide 200 mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7789, ANCOVA; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.61 to 0.81]

4. Secondary Outcome: Change From Baseline Over 2 Weeks in Participant-Reported Morning and Evening Instantaneous Total Ocular Symptom Scores
Description: The instantaneous TOSS is defined as the sum of the participant-rated instantaneous symptom scores for 3 ocular symptoms of itching/burning eyes, tearing/watering eyes, and redness of eyes at the time of evaluation. Each symptom was evaluated by the participant in an assessment diary, once in the morning (AM score) and after 12 hours in the evening (PM score) over 2 weeks of treatment period and was rated on a severity scale ranging from 0 to 3, where: 0 = absent, 1 = mild, 2 = moderate, and 3 = severe (symptom hard to tolerate, interferes with daily activities/sleeping). Instantaneous TOSS score ranges from 0-9 with 0 representing an absence of symptoms and 9 representing severe symptoms. The baseline value was defined as the average score over the Day -6 to Day 0. Change from Baseline was thus calculated as the 2-week average score recorded from Day 1 up to Day 14 minus the Baseline score.
Time Frame: Baseline and Week 1 up to Week 2 (entire treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ciclesonide 200 mcg | Placebo
Number analyzed (Participants) | 40 | 40
scores on a scale
  Baseline | 4.74 (1.25) | 4.69 (1.53)
  Change Over 2 Weeks | -1.56 (1.67) | -1.61 (1.73)
Statistical Analysis 1: Comparison: Ciclesonide 200 mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6630, ANCOVA; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.55 to 0.86]

5. Secondary Outcome: Change From Baseline Over 2 Weeks in Participant-Reported Individual Morning and Evening Reflective Total Nasal Symptom Score
Description: as for outcome 1
Time Frame: Baseline and Week 1 up to Week 2 (entire treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ciclesonide 200 mcg | Placebo
Number analyzed (Participants) | 40 | 40
scores on a scale
  Nasal Congestion: Baseline | 2.19 (0.50) | 2.22 (0.38)
  Nasal Congestion: Change Over 2 Weeks | -0.70 (0.64) | -0.62 (0.63)
  Runny nose: Baseline | 2.04 (0.61) | 2.01 (0.64)
  Runny nose: Change Over 2 Weeks | -0.79 (0.71) | -0.77 (0.64)
  Itchy Nose: Baseline | 1.77 (0.65) | 1.76 (0.43)
  Itchy Nose: Change Over 2 Weeks | -0.64 (0.66) | -0.64 (0.58)
  Sneezing: Baseline | 1.80 (0.58) | 1.73 (0.56)
  Sneezing: Change Over 2 Weeks | -0.71 (0.76) | -0.64 (0.69)
Statistical Analysis 1: Comparison: Ciclesonide 200 mcg vs Placebo; Nasal congestion: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.5593, ANCOVA; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.35 to 0.19]
Statistical Analysis 2: Comparison: Ciclesonide 200 mcg vs Placebo; Runny nose: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.7085, ANCOVA; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.22 to 0.33]
Statistical Analysis 3: Comparison: Ciclesonide 200 mcg vs Placebo; Itching: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.7309, ANCOVA; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.22 to 0.31]
Statistical Analysis 4: Comparison: Ciclesonide 200 mcg vs Placebo; Sneezing: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.9584, ANCOVA; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.29 to 0.30]

6. Secondary Outcome: Change From Baseline Over 2 Weeks in Participant-Reported Individual Morning and Evening Reflective Total Ocular Symptom Score
Description: as for outcome 3
Time Frame: Baseline and Week 1 up to Week 2 (entire treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ciclesonide 200 mcg | Placebo
Number analyzed (Participants) | 40 | 40
scores on a scale
  Itching/Burning Eyes: Baseline | 1.85 (0.54) | 1.79 (0.53)
  Itching/Burning Eyes: Change Over 2 Weeks | -0.63 (0.77) | -0.73 (0.68)
  Redness: Baseline | 1.57 (0.63) | 1.67 (0.53)
  Redness: Change Over 2 Weeks | -0.59 (0.59) | -0.52 (0.64)
  Tearing/Watering Eyes: Baseline | 1.37 (0.53) | 1.29 (0.58)
  Tearing/Watering Eyes: Change Over 2 Weeks | -0.45 (0.56) | -0.43 (0.61)
Statistical Analysis 1: Comparison: Ciclesonide 200 mcg vs Placebo; Itching/Burning Eyes: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.2266, ANCOVA; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.11 to 0.46]
Statistical Analysis 2: Comparison: Ciclesonide 200 mcg vs Placebo; Redness: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.4888, ANCOVA; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.35 to 0.17]
Statistical Analysis 3: Comparison: Ciclesonide 200 mcg vs Placebo; Tearing/Watering Eyes: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.8316, ANCOVA; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.22 to 0.27]

7. Secondary Outcome: Change From Baseline Over 2 Weeks in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Total Score
Description: The RQLQ is a 28-item, disease-specific quality of life questionnaire that measures the functional (physical, emotional, and social) problems troublesome to adults with allergies. The RQLQ has 28 questions in 7 domains (activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms and emotional). All 28 questions were evaluated by the participant in an assessment diary over 2 weeks of treatment period and was rated on a 7-point severity scale ranging from 0 to 6, where 0 = least severe to 6 = extremely severe. Overall total score was calculated by taking the mean of the response of all individual 28 questions. The baseline value was defined as the average score over the Day -6 to Day 0. Change from Baseline was thus calculated as the 2-week average score recorded from Day 1 up to Day 14 minus the Baseline score.
Time Frame: Baseline and Week 1 up to Week 2 (entire treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ciclesonide 200 mcg | Placebo
Number analyzed (Participants) | 40 | 40
scores on a scale
  Baseline | 3.31 (0.83) | 3.24 (0.85)
  Change Over 2 Weeks | -1.40 (1.26) | -1.09 (1.08)
Statistical Analysis 1: Comparison: Ciclesonide 200 mcg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2968, ANCOVA; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.80 to 0.25]

8. Secondary Outcome: Change From Baseline Over 2 Weeks in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Individual Domain Score
Description: The RQLQ is a 28-item, disease-specific quality of life questionnaire that measures the functional (physical, emotional, and social) problems troublesome to adults with allergies. The RQLQ has 28 questions in 7 domains (activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms and emotional). All 28 questions were evaluated by the participant in an assessment diary over 2 weeks of treatment period and was rated on a 7-point severity scale ranging from 0 to 6, where 0 = least severe to 6 = extremely severe. Overall domain scores were calculated by taking the mean of the response of the relevant questions. The baseline value was defined as the average score over the Day -6 to Day 0. Change from Baseline was thus calculated as the 2-week average score recorded from Day 1 up to Day 14 minus the Baseline score.
Time Frame: Baseline and Week 1 up to Week 2 (entire treatment period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ciclesonide 200 mcg | Placebo
Number analyzed (Participants) | 40 | 40
scores on a scale
  Activities: Baseline | 4.07 (0.77) | 4.05 (1.03)
  Activities: Change Over 2 Weeks | -1.55 (1.31) | -1.24 (1.23)
  Sleep: Baseline | 3.22 (1.41) | 3.15 (1.31)
  Sleep: Change Over 2 Weeks | -1.38 (1.52) | -1.02 (1.39)
  Non-Nose/Eye Symptoms: Baseline | 2.74 (1.21) | 2.85 (1.00)
  Non-Nose/Eye Symptoms: Change Over 2 Weeks | -1.07 (1.23) | -0.90 (1.04)
  Practical Problems: Baseline | 4.01 (1.07) | 3.50 (1.25)
  Practical Problems: Change Over 2 Weeks | -1.76 (1.58) | -1.18 (1.26)
  Nasal Symptoms: Baseline | 4.05 (0.94) | 3.90 (1.19)
  Nasal Symptoms: Change Over 2 Weeks | -1.78 (1.67) | -1.44 (1.45)
  Eye Symptoms: Baseline | 3.01 (1.19) | 2.91 (1.07)
  Eye Symptoms: Change Over 2 Weeks | -1.28 (1.40) | -1.03 (1.14)
  Emotional: Baseline | 2.82 (1.35) | 2.89 (1.18)
  Emotional: Change Over 2 Weeks | -1.39 (1.45) | -1.06 (1.44)
Statistical Analysis 1: Comparison: Ciclesonide 200 mcg vs Placebo; Activities: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.3533, ANCOVA; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.85 to 0.31]
Statistical Analysis 2: Comparison: Ciclesonide 200 mcg vs Placebo; Sleep: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.3712, ANCOVA; Mean Difference (Net) = -0.26, 95% CI 2-sided [-0.84 to 0.32]
Statistical Analysis 3: Comparison: Ciclesonide 200 mcg vs Placebo; Non-nose/Eye symptoms: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.4098, ANCOVA; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.69 to 0.29]
Statistical Analysis 4: Comparison: Ciclesonide 200 mcg vs Placebo; Practical Problems: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.2683, ANCOVA; Mean Difference (Net) = -0.36, 95% CI 2-sided [-1.00 to 0.28]
Statistical Analysis 5: Comparison: Ciclesonide 200 mcg vs Placebo; Nasal Symptoms: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.4643, ANCOVA; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.82 to 0.38]
Statistical Analysis 6: Comparison: Ciclesonide 200 mcg vs Placebo; Eye symptoms: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.4502, ANCOVA; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.74 to 0.33]
Statistical Analysis 7: Comparison: Ciclesonide 200 mcg vs Placebo; Emotional: An ANCOVA model adjusted for treatment, site and the baseline score was used to test a null hypothesis of no difference between the treatment groups against a two-sided alternative hypothesis at the 5% level of significance; Test type: Superiority or Other; p = 0.1770, ANCOVA; Mean Difference (Net) = -0.39, 95% CI 2-sided [-0.95 to 0.18]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days after the last dose of double-blind study drug (Day 29).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ciclesonide 200 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 6/40 | 10/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciclesonide 200 mcg (N=40) | Placebo (N=40)
Insomnia (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 6
Migraine (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Decreased activity (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.